CLINICAL TRIAL: NCT01747213
Title: Phase I, Double-Blind, Placebo-Controlled, Ascending, Single-Dose, Safety, Tolerability and Pharmacokinetic Study of Bisnorcymserine (BNC), a Highly Selective Inhibitor of Butyrylcholinesterase, in Healthy Adult Volunteers
Brief Title: Bisnorcymserine in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 130034; 13-AG-0034
Record Dates: First submitted 2012-12-08; First posted 2012-12-11 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-04-18

CONDITIONS: Healthy Volunteers
Keywords: Clinical Trial; Alzheimer Disease; Healthy Volunteers; Neurotransmitters
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BNC (Experimental): Bisnorcymserine tartrate
  Interventions: Drug: BNC
- Placebo (Placebo Comparator): microcrystalline celluose
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BNC
  Arms: BNC
Other: Placebo — Microcrystalline cellulose fiber
  Arms: Placebo

SUMMARY:
Background:

- Alzheimer s disease (AD) is a brain disease that impairs memory, cognitive abilities and the ability to function independently. It is the most common cause of dementia in older people. It is caused by abnormal proteins in the brain that affect how neurons communicate with each other. Researchers are looking for drugs that can slow down the disease or treat its symptoms. One drug, called bisnorcymserine (BNC), may help improve brain function and symptoms in people with AD. BNC is designed to block a chemical that affects how neurons communicate with each other. Researchers want to see how BNC works in healthy older volunteers.

Objectives:

- To look at how the body processes bisnorcymserine taken by mouth and how safe it is for healthy older volunteers.

Eligibility:

- Healthy volunteers at least 55 years of age.

Design:

* Participants will be screened with a physical exam, medical history, and blood and urine tests.
* Within 3 weeks from the screening visit, participants will come to the National Institute on Aging clinical unit for a 2-night stay. On the morning of the second day, they will take either a BNC capsule or a placebo. They will not know which tablet they are taking.
* Blood samples will be collected frequently throughout the second and third days of the study visit. The last blood sample will be collected about 32 hours after taking the study capsule. Participants will have heart function tests and other exams during the visit. Once the tests are done, they will leave the clinical center.
* Participants will have a final follow-up visit about 1 week after leaving the clinical center.

DETAILED DESCRIPTION:
Objective: Alzheimer s disease (AD) is a progressive neurodegenerative disease that impairs memory and other cognitive abilities, as well as behavior and the ability to function independently. It is the most common cause of dementia among older people. Alzheimer s disease is characterized by deficits in several neurotransmitter systems, most prominently acetylcholine (Ach). The cholinergic deficit in the AD brain is associated with the cognitive and functional symptoms in AD. Restoring this deficit in the cholinergic system is one proven approach for symptomatic treatment in AD. The action of Ach in the brain is terminated mainly by two enzymes called cholinesterases (ChEs): acetylcholinesterase (AChE) and butyrylcholinesterase (BChE). Inhibitors of these enzymes therefore augment the activity of surviving Ach neurons in AD. All ChEs inhibitors currently approved for the treatment of AD mainly inhibit AChE and, secondarily and to a varying extent, BChE. Reversible and brain-specific BChE inhibitors have been developed as a class of drugs called cymserine analogs. Scientists at the NIA/NIH have developed a novel BChE inhibitor called Bisnorcymserine (BNC). Pre-clinical evidence suggests that BNC may be a safe treatment for Alzheimer s disease. Based on this, we propose this first-in-human study to evaluate the safety, tolerability and pharmacokinetics of single doses of BNC tartrate administered orally.

Study population: Healthy volunteers aged 55 years and older.

Design: Double blind placebo-controlled Phase I clinical Trial of single oral doses of BNC doses in an ascending schedule: 20, 40mg, 80 mg, 120 mg, 160 mg, 270 mg and 380 mg. Each dose will be tested in groups of 8 subjects. Six subjects in each cohort will receive active drug and two will receive placebo. Subjects will be kept in the unit and followed clinically and with laboratory tests for adverse effects for 32 hours; they will return for a follow-up visit to assess safety in about 7 days. A Data Safety Monitoring Board will evaluate the safety and tolerability associated with each dose level before the next higher dose is tested in a new cohort. All research will be performed at the National Institute on Aging (NIA) Clinical Research Unit located on the 5th floor of MedStar Harbor Hospital.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age greater than or equal to 55 years.
* Mini Mental State Examination (MMSE) > 27 at screening and at Visit 2-Day 1.
* Women who are able to become pregnant must have a negative urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) at screening and prior to study drug administration
* Both men who are able to father children and women of childbearing potential must be willing to use an adequate method of contraception (see section 7) to avoid conception throughout the study and for up to 30 days of study drug administration.
* Body mass index (BMI) of 18.5 to 34.0, inclusive, and a total body weight of > 50 kg (110 pounds).
* Participants should be in good general physical and mental health as determined by medical history, a baseline physical examination, vital signs, clinical laboratory tests and electrocardiogram (EKG). Participants may have common age-related disorders (such as hypertension, type II diabetes, dyslipidemia, hypothyroidism) as long as these disorders are under good control by diet or medications.
* Able to sign own consent

EXCLUSION CRITERIA:

* Any clinically significant medical and psychiatric condition (including asthma active within the last 10 years or COPD, and drug abuse and dependency).
* Subject has used any tobacco products in the past 3 months.
* A history of significant allergy to any drug or systemic allergic disease (e.g., urticaria, atopic dermatitis).
* Pregnant or lactating females.
* Subject with a positive urine test for drugs of abuse at screening or at admission to the clinic on study Day 1.
* Subject has consumed any alcohol within 48 hours prior to Visit 2; and cannot or is unwilling, thereafter to abstain from drinking alcohol for the remainder of the subject s study participation.
* Subject is positive for HIV, hepatitis B surface antigen or hepatitis C antibody tests at screening.
* Any clinically significant laboratory abnormality. These include:

  * CBC: WBC < 3000 /mm^3; Hb < 12 g/dL; Liver function tests: ALT, AST, Bilirubin (total, direct, indirect), Alkaline Phosphatase > 1.5 x the upper normal limit of the laboratory
  * Serum Creatinine > 1.5 mg/dL; Serum Glucose >150mg/dL
  * Resting supine blood pressure outside of a systolic blood pressure range of 90-140 mmHg or a diastolic blood pressure outside a range of 50-90 mmHg on two consecutive measurements taken up to 10 minutes apart.Resting supine heart rate greater than 100 bpm or less than or equal to 55 55 bpm on two consecutive measurements taken up to 10 minutes apart.
  * Any clinically significant abnormality on screening 12-lead EKG (e.g., heart block, conduction disorders, ventricular and/or atrial arrhythmias).
* Routine or PRN consumption of the following herbal/dietary supplements are not permitted, if used within 2 weeks before the screening visit at doses higher than the recommended daily intake: Omega-3 fatty acids (> 1000 mg/day), Vitamin E (> 400IU/day). Ginkgo biloba, St. John's wort and ginseng are not permitted, if used at any dose within 2 weeks before the screening visit.
* Medications that are excluded are:

  * Insulin
  * Anti-parkinsonian medications (such as levodopa/carbidopa, amantadine, bromocriptine, pergolide, selegiline)
  * Typical or atypical neuroleptics
  * Narcotic analgesics at any dose within 4 weeks prior to screening.
  * Long-acting benzodiazepines or barbiturates (such as clonazepam, diazepam, phenobarbital) within 4 weeks prior to screening
  * Short-acting anxiolytics or sedative hypnotics more frequently than 2 times per week within 4 weeks prior to screening (sedative hypnotics should not be used within 102 hours of study drug administration)
  * Medications with known significant cholinergic or anticholinergic side effects (such as pyridostigmine, tricyclic antidepressants, meclizine, oxybutynin) within 4 weeks prior to screening
  * Anti-convulsants (such as phenytoin, Phenobarbital, carbamazepine) within 2 months prior to screening
  * Medications for Alzheimer s disease (such as donepezil or memantine)
  * Beta-Blockers
  * Corticosteroids (Systemic)
  * Neuromuscular-Blocking Agents (non-depolarizing)
  * Succinylcholine
  * Any other drug (including prescription, over the counter medications and supplements) that may pose a risk to the subject or produce overlapping side effects with the study medication. Participants will not be taken off of medications for the purpose of this study.
* Donation or loss of 400 mL or more of blood within 56 days prior to and subsequent to screening.
* Participation in another research study involving an investigational drug within 30 days or 5 half-lives, whichever is longer.
* Known allergy or hypersensitivity to the investigational study drug and to the microcrystalline cellulose used as placebo.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-01-29 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | Will be completed in one year
  Safety and tolerability will be determined based on the frequency of AEs of any grade in BNC and placebo groups. AEs will be determined based on clinical symptoms and signs, vital signs, safety laboratory tests, EKG and continuous cardiac monitoring, MMSE, and C-SSRS.

SECONDARY OUTCOMES:
pharmacokinetic profile (parameters) | Will be completed in one year
  The pharmacokinetic profile of a single oral dose of BNC in a capsule will be determined, including evaluation of AUC, Tmax, Cmax, elimination rate constant, T1/2, clearance and volume of distribution. In addition, we will measure pharmacodynamics parameters, including acetyl-cholinesterase and butyryl-cholinesterase activity

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios I Kapogiannis, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (2):
- United States (2):
  - National Institute on Aging, Clinical Research Unit, Baltimore, Maryland
  - Harbor Hospital Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Undecided
There is ongoing discussion within the NIA IRP and a plan has not been finalized yet.

REFERENCES:
- [Background] Arendt T, Bigl V, Walther F, Sonntag M. Decreased ratio of CSF acetylcholinesterase to butyrylcholinesterase activity in Alzheimer's disease. Lancet. 1984 Jan 21;1(8369):173. doi: 10.1016/s0140-6736(84)90116-8. No abstract available. PMID 6140490
- [Background] Cummings JL. Use of cholinesterase inhibitors in clinical practice: evidence-based recommendations. Am J Geriatr Psychiatry. 2003 Mar-Apr;11(2):131-45. PMID 12611743
- [Background] Darvesh S, Grantham DL, Hopkins DA. Distribution of butyrylcholinesterase in the human amygdala and hippocampal formation. J Comp Neurol. 1998 Apr 13;393(3):374-90. PMID 9548556
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-AG-0034.html